CLINICAL TRIAL: NCT03035825
Title: A Randomized Controlled Trial for Efficacy of Oral Moisturizing Jelly on Oral Health and Nutrition in Post-radiotherapy Head and Neck Cancer Patients With Xerostomia
Brief Title: Efficacy of Oral Moisturizing Jelly on Oral Health and Nutrition in Post-radiotherapy Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dental Innovation Foundation Under Royal Patronage (Other)
Collaborators: Mahidol University (Other); Srinakharinwirot University (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DIF-05
Record Dates: First submitted 2017-01-25; First posted 2017-01-30 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Cancer of Head Neck; Radiation-Induced Xerostomia; Dry Mouth
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia | interventions — Saliva, Artificial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Moisturizing Jelly (Experimental): Daily intake of oral moisturizing jelly 5 times/day for two months
  Interventions: Dietary Supplement: Oral moisturizing jelly
- Artificial saliva (Active Comparator): Daily use of non-edible oral lubricating gel 5 times/day for two months
  Interventions: Other: Artificial saliva

INTERVENTIONS:
Dietary Supplement: Oral moisturizing jelly — Gel-based artificial saliva is an edible non-nutritious gel intended to relieve dry mouth
  Arms: Oral Moisturizing Jelly
Other: Artificial saliva — A non-edible oral lubricating gel for dry mouth patients
  Other Names: Dry mouth gel
  Arms: Artificial saliva

SUMMARY:
This randomized control trial aims to investigate the efficacy of oral moisturizing jelly in head and neck cancer patients with xerostomia.

DETAILED DESCRIPTION:
Oral moisturizing jelly is a novel edible, gel-based artificial saliva. It has been proven effective in reducing dry mouth sign and symptoms in elderly patients with xerostomia. This randomized control trial intends to determine if continuous use of oral moisturizing jelly may be effective in reduction of signs and symptoms of dry mouth, improvement of biochemical properties of saliva, subjective swallow ability, appetite, tolerance to spicy food, energy intake and reduce umami taste recognition threshold.

ELIGIBILITY:
Inclusion Criteria:

1. Xerostomic head and neck cancer patients who finish radiotherapy for at least 1 month.
2. If undergoing chemotherapy, have to finish for at least 2 weeks.
3. Have subjective dry mouth scores at least 3
4. Can perform oral intake without aspiration
5. Can communicate well

Exclusion Criteria:

1. Has recurrence of cancer
2. Has mucositis more than grade 1
3. Has oral infection such as candidiasis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in subjective dry mouth score compared to baseline | Baseline, 1 and 2 months after intervention
  Evaluation of subjective dry mouth score by questionaire

SECONDARY OUTCOMES:
Changes in objective dry mouth score compared to baseline | Baseline, 1 and 2 months after intervention
  Evaluation of objective dry mouth score by oral examination
Changes in salivary pH compared to baseline | Baseline, 1 and 2 months after intervention
  Evaluation of salivary pH using pH indicator paper
Changes in salivary buffering capacity compared to baseline | Baseline, 1 and 2 months after intervention
  Evaluation of salivary buffering capacity using a commercial saliva check buffer kit
Changes in Candidal counts of saliva compared to baseline | Baseline, 1 and 2 months after intervention
  Evaluation of number of fungal colonies of Candida spp. in saliva by culture
Changes in energy intake compared to baseline | Baseline, 1 and 2 months after intervention
  Evaluation of energy intake per day using dietary record and analysis
Changes in subjective swallow ability compared to baseline | Baseline, 1 and 2 months after intervention
  Evaluation of subjective swallow ability using EAT-10 questionaire
Changes in appetite compared to baseline | Baseline, 1 and 2 months after intervention
  Evaluation of appetite using questionnaire
Changes in tolerance to spicy food | Baseline, 1 and 2 months after intervention
  Evaluation of tolerance to spicy food using questionnaire
Changes in umami taste recognition threshold compared to baseline | Baseline, 1 and 2 months after intervention
  Evaluation of umami taste recognition threshold using filter paper disc method

CONTACTS AND LOCATIONS:
Overall Officials: Aroonwan Lam-ubol, DDS, PhD, Principal Investigator — Srinakarinwirot University
Locations (1):
- Chonburi Cancer Hospital, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam-Ubol A, Matangkasombut O, Trachootham D, Tarapan S, Sattabanasuk V, Talungchit S, Paemuang W, Phonyiam T, Chokchaitam O, Mungkung OO. Efficacy of gel-based artificial saliva on Candida colonization and saliva properties in xerostomic post-radiotherapy head and neck cancer patients: a randomized controlled trial. Clin Oral Investig. 2021 Apr;25(4):1815-1827. doi: 10.1007/s00784-020-03484-1. Epub 2020 Aug 10. PMID 32779011
- [Derived] Nuchit S, Lam-Ubol A, Paemuang W, Talungchit S, Chokchaitam O, Mungkung OO, Pongcharoen T, Trachootham D. Alleviation of dry mouth by saliva substitutes improved swallowing ability and clinical nutritional status of post-radiotherapy head and neck cancer patients: a randomized controlled trial. Support Care Cancer. 2020 Jun;28(6):2817-2828. doi: 10.1007/s00520-019-05132-1. Epub 2019 Nov 15. PMID 31732852